CLINICAL TRIAL: NCT00096551
Title: A Phase I Feasibility Study of an Intraprostatic PSA-Based Vaccine in Men With Prostate Cancer and Local Failure Following Radiotherapy or Cryotherapy or Clinical Progression on Androgen Deprivation Therapy in the Absence of Local Definitive Therapy
Brief Title: A Phase I Feasibility Study of an Intraprostatic PSA-Based Vaccine in Men With Prostate Cancer With Local Failure Following Radiotherapy or Cryotherapy or Clinical Progression on Androgen Deprivation Therapy in the Absence of Local Definitive Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050017; 05-C-0017; NCT00098449 (obsolete NCT alias)
Record Dates: First submitted 2006-07-07; First posted 2004-11-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-25

CONDITIONS: Prostatic Neoplasms
Keywords: Biochemical Failure; Immunotherapy; TRICOM; Pox-virus; Fowlpox; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Fowlpox

INTERVENTIONS:
Drug: Recombinant Vaccinia-PSA(L155)/TRICOM (PROSTVAC-V/TRICOM)
Drug: Recombinant Fowlpox-PSA(L155)/TRICOM (PROSTVAC-F/TRICOM)
Drug: Recombinant Fowlpox-GM-CSF

SUMMARY:
Background:

* Pox viral vectors can induce a PSA-specific T-cell responses and clinical responses in patients with advanced prostate cancer.
* Intratumoral vaccines of recombinant fowlpox vectors appear to be more potent in inducing antitumor effects than the s.c. route of administration, especially when the recombinant rF-vector given intratumorally is preceded by a rV-recombinant given s.c. This may be due to:
* Making the tumor cell an antigen presenting cell via upregulation of both antigen (signal 1) and costimulatory molecules (signal 2).
* Making the tumor cell more susceptible to killing via upregulation of ICAM.
* The increased expression of perforin in peptide-specific T cells that came into contact with the TRICOM-infected targets.
* Potentially allowing the immune system to select for other tumor encoded antigens to generate a polyvalent immune response.

Objectives:

* 1: Safety and feasibility of an intraprostatic vaccine strategy.
* 2: To assess the change in PSA-specific T-cell response as measured by ELISPOT assay.
* 2: To evaluate T-cell infiltration histologically in patients who have pre- and post-vaccine prostate biopsies.

Eligibility:

* Must have either a) biopsy proven, locally recurrent prostate cancer following local radiation as defined by the ASTRO consensus criteria as 3 consecutively rising PSA levels or b) have refused or not be candidates for local definitive therapy (surgery or radiation therapy) and have clinically progressive disease on androgen deprivation therapy (eg. three increases in PSA over nadir, separated by at least one week). For patients with previous RT, the biopsy confirming local recurrence must be done at least 18 months after the completion of RT.
* Since this may also generate a systemic immune response, patients with minimal extraprostatic disease may be enrolled.
* Hepatic function: Bilirubin < 1.5 mg/dl, AST and ALT< 2.5 times upper limit of normal

Design:

* Dose escalation Phase I design. Each cohort will consist of 3-6 patients, with cohorts 4 & 5 restricted to include only HLA-A2 + patients; maximum accrual is 30
* Patients in all cohorts receive initial priming with rV- PSA(L155)/TRICOM and rF-GM-CSF s.c.
* The first two cohorts utilize a booster intraprostatic with dose escalation of rF-PSA(L155)/TRICOM.
* Third and fourth cohorts add dose escalations of rF-GM-CSF along with the highest dose of rF-PSA(L155)/TRICOM
* Last (5th) cohort u...

DETAILED DESCRIPTION:
Background:

* Pox viral vectors can induce a PSA-specific T-cell responses and clinical responses in patients with advanced prostate cancer.
* Intratumoral vaccines of recombinant fowlpox vectors appear to be more potent in inducing antitumor effects than the s.c. route of administration, especially when the recombinant rF-vector given intratumorally is preceded by a rV-recombinant given s.c. This may be due to:
* Making the tumor cell an antigen presenting cell via upregulation of both antigen (signal 1) and costimulatory molecules (signal 2).
* Making the tumor cell more susceptible to killing via upregulation of ICAM.
* The increased expression of perforin in peptide-specific T cells that came into contact with the TRICOM-infected targets.
* Potentially allowing the immune system to select for other tumor encoded antigens to generate a polyvalent immune response.

Objectives:

* 1: Safety and feasibility of an intraprostatic vaccine strategy.
* 2: To assess the change in PSA-specific T-cell response as measured by ELISPOT assay.
* 2: To evaluate T-cell infiltration histologically in patients who have pre- and post-vaccine prostate biopsies.

Eligibility:

* Must have either a) biopsy proven, locally recurrent prostate cancer following local radiation as defined by the ASTRO consensus criteria as 3 consecutively rising PSA levels or b) have refused or not be candidates for local definitive therapy (surgery or radiation therapy) and have clinically progressive disease on androgen deprivation therapy (eg. three increases in PSA over nadir, separated by at least one week). For patients with previous RT, the biopsy confirming local recurrence must be done at least 18 months after the completion of RT.
* Since this may also generate a systemic immune response, patients with minimal extraprostatic disease may be enrolled.
* Hepatic function: Bilirubin less than 1.5 mg/dl, AST and ALT less than 2.5 times upper limit of normal.

Design:

* Dose escalation Phase I design. Each cohort will consist of 3-6 patients; maximum accrual is 30
* Patients in all cohorts receive initial priming with rV- PSA(L155)/TRICOM and rF-GM-CSF s.c.
* The first two cohorts utilize a booster intraprostatic with dose escalation of rF-PSA(L155)/TRICOM.
* Third and fourth cohorts add dose escalations of rF-GM-CSF along with the highest dose of rF-PSA(L155)/TRICOM.
* Last (5th) cohort utilizes booster intraprostatic vaccine (rF-PSA(L155)/TRICOM and rF-GM-CSF) with simultaneous identical booster vaccine given s.c.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology at: NIH Clinical Center, National Institutes of Health (NIH), the National Naval Medical Center, or Walter Reed Army Medical Center prior to starting this study. If no pathologic specimen is available, patients may enroll with a pathologist's report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

B. Must have either a) biopsy proven, locally recurrent prostate cancer following local radiation or cyrotherapy as defined by the ASTRO consensus criteria as 3 consecutively rising PSA levels or b) have refused or not be candidates for local definitive therapy (surgery or radiation therapy) and have clinically progressive disease on androgen deprivation therapy (e.g., three increases in PSA over nadir, separated by at least one week). For patients with previous RT, the biopsy confirming local recurrence must be done at least 18 months after the completion of RT.

Since this may also generate a systemic immune response, patients with minimal extraprostatic disease may be enrolled.

C. Agree to use adequate contraception prior to study entry and for at least 4 months following the last vaccine injection.

D. Life expectancy greater than or equal to 6 months.

E. ECOG performance status of 0 to 2 (see Appendix A).

F. Recovered from any acute toxicity related to prior therapy, including surgery, and radiation (treatment must have been completed at least 4 weeks prior to being eligible for the study).

G. Hematological eligibility parameters (within 16 days of starting therapy, see Appendix D).

Granulocyte count greater than or equal to 1,500/mm3

Platelet count greater than or equal to 100,000/mm3

Lymphocyte count greater than or equal to 500/mm3

Hgb greater than or equal to 10 Gm/dL

H. Biochemical eligibility parameters (within 16 days of starting therapy):

-A 24-hour urine collection for baseline to measure creatinine clearance, protein and electrolytes. CrCl greater than 60mL/min, proteinuria less than 1000 milligrams per 24 hours, and no abnormal sediment. Serum creatinine not above normal limits OR creatinine clearance on a 24 hour urine collection of greater than 60 mL/min. For patients who are not able to obtain an accurate collection, a calculated creatinine clearance and urine analysis for protein may be used. Any abnormalities in the sediment or the presence of hematuria without a likely underlying cause should prompt the investigator to consider an evaluation by a nephrologist or urologist for evidence of underlying renal pathology.

Patients may be eligible if the underlying cause of the abnormality is determined to be non-renal.

-Hepatic function: Bilirubin equal to 1.5 mg/dL or patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 mg/dL, AST and ALT less than 2.5 times upper limit of normal.

I. No other active malignancies within the past 12 months (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder) or life threatening illnesses.

J. Willing to travel to the NIH for follow-up visits.

K. 18 years of age or greater.

L. Vaccinia-naive or vaccinia immune.

M. Able to understand and sign informed consent.

N. Tested for HLA-A2; however, the results of this test will not affect entry into this study. This test may be drawn by the patient's referring physician at the time of referral (see Screening Consent for HLA typing). This consent will be mailed to the patient and discussed with patient. The signed consent will be signed with a non-family member witness and then mailed to the assigned research nurse at the NIH Clinical Center.

O. Concurrent hormonal therapy will be allowed.

P. PT / PTT will be drawn prior to any invasive protocol related procedure (i.e., prostate biopsy or intraprostatic injection) and standard clinical guidelines followed.

EXCLUSION CRITERIA:

A. Patients should have no evidence of being immunocompromised as listed below.

* Human immunodeficiency virus positivity due to the potential for decreased tolerance and may be at risk for severe side effects.
* Active autoimmune diseases such as, Addison's disease, Hashimoto's thyroiditis, or systemic lupus erythematous, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome active Grave's disease. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including CNS, heart, lungs, kidneys, skin, and GI tract will be allowed.
* Hepatitis B or C positivity.
* Concurrent use of systemic steroids, except for physiologic doses for systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Steroid eye drops are contraindicated for at least 2 weeks prior vaccinia vaccination and at least 4 weeks post vaccinia vaccination.

B. History of allergy or untoward reaction to prior vaccination with vaccinia virus or to any component of the vaccinia vaccine regimen.

C. Must be able to avoid close household contact (close household contacts are those who share housing or have close physical contact) for at least three weeks after recombinant vaccinia vaccination with persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection.

D. Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.

E. Patients with cardiac disease that have fatigue, palpitation, dyspnea or angina with ordinary physical activity (New York Heart Association class 2 or greater) are not eligible.

F. Patients who have objective evidence of congestive heart failure by physical exam or imaging are not eligible.

G. Patients with pulmonary disease that have fatigue or dyspnea with ordinary physical activity are not eligible.

H. Concurrent chemotherapy.

I. Clinically active brain metastasis, or with a history of seizures, encephalitis, or multiple sclerosis.

J. Serious hypersensitivity reaction to egg products.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-11-01; Primary Completion 2009-12-11 (Actual); Study Completion 2011-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lattouf JB, Arlen PM, Pinto PA, Gulley JL. A phase I feasibility study of an intraprostatic prostate-specific antigen-based vaccine in patients with prostate cancer with local failure after radiation therapy or clinical progression on androgen-deprivation therapy in the absence of local definitive therapy. Clin Genitourin Cancer. 2006 Jun;5(1):89-92. doi: 10.3816/CGC.2006.n.024. No abstract available. PMID 16859586
- [Background] Kudo-Saito C, Schlom J, Hodge JW. Intratumoral vaccination and diversified subcutaneous/ intratumoral vaccination with recombinant poxviruses encoding a tumor antigen and multiple costimulatory molecules. Clin Cancer Res. 2004 Feb 1;10(3):1090-9. doi: 10.1158/1078-0432.ccr-03-0145. PMID 14871989